CLINICAL TRIAL: NCT05390749
Title: Sequential Treatment Regimens With RO-MTX After Pomalidomide, Orelabrutinib, Rituximab (POR) as Frontline Therapy for Primary Central Nervous System Lymphoma: a Multicenter Prospective Single Arm Trial
Brief Title: Sequential Treatment With RO-MTX After Pomalidomide, Orelabrutinib, Rituximab (POR) in Newly-diagnosed PCNSL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-013
Record Dates: First submitted 2022-05-11; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Orelabrutinib; Pomalidomide; Rituximab; primary central nervous system lymphoma; methotrexate
MeSH Terms: interventions — orelabrutinib; pomalidomide; Rituximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POR-ROMTX (Experimental): The experimental arm will be treated with 4 cycles of POR regimen （Pomalidomide 4mg d1-d14, Orelabrutinib 150mg d1-d21, Rituximab 375mg/m2 d1, 21 days per cycle). The response will be evaluated every 2 cycles. The patients with PD will drop out of the study.Patients with CR/PR/SD after 4 cycles of POR treatment will be treated with 2 cycles of RO-MTX regimen（methotrexate 3.5g/m2 civ d1, Orelabrutinib 150mg d1-d21, Rituximab 375mg/m2 d1, 21 days per cycle).
  Interventions: Drug: Orelabrutinib; Drug: Pomalidomide; Drug: Rituximab; Drug: Methotrexate

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib will be given as 150mg orally d1-d21 for 6 cycles,every 21 days for 1 cycle.
Drug: Pomalidomide — Pomalidomide will be given as 4mg d1-d14 for 4 cycles,every 21 days for 1 cycle.
Drug: Rituximab — Rituximab 375mg/m2 intravenous infusion d1, every 21 days for 1 cycle. 6 cycles will be prescribed as protocol
Drug: Methotrexate — methotrexate 3.5g/m2 civ d1/cycle5-6

SUMMARY:
This is a multicenter prospective single arm phase II study, and the purpose of this study is to evaluate the safety and efficacy of sequential treatment regimens with RO-MTX after pomalidomide, orelabrutinib, rituximab (POR) in newly-diagnosed primary central nervous system lymphoma, and explore the feasibility of chemo-free treatment in PCNSL. The primary objective was the overall response rate (ORR; defined as partial response [PR] or better) after 4 cycles of POR.

DETAILED DESCRIPTION:
There are 2 sections of this trial. Step1: the patients will be treated with 4 cycles of POR regimen （Pomalidomide 4mg d1-d14, Orelabrutinib 150mg d1-d21, Rituximab 375mg/m2 d1, 21 days per cycle). The response will be evaluated every 2 cycles. The patients with PD will drop out of the study. Step2: Patients with CR/PR/SD after 4 cycles of POR treatment will be treated with 2 cycles of RO-MTX regimen（methotrexate 3.5g/m2 civ d1, Orelabrutinib 150mg d1-d21, Rituximab 375mg/m2 d1, 21 days per cycle). After 6 cycles of induction therapy, all patients were followed for survival data every 12 week until disease progression, disease recurrence, death, or study termination. Patients with progression were also followed up for survival data as above. Overall survival will be followed up to 3 years after the last subject entered the study. Establishing the feasibility of chemo-free treatment in primary central nervous system lymphoma will provide the foundation for a larger study of efficacy and long-term outcomes of chemo-free therapy for patients with PCNSL.

ELIGIBILITY:
Inclusion Criteria:

* • Newly diagnosed primary central nervous system lymphoma

  * Pathological type is B cell lymphoma
  * Age 18-70 years
  * Demonstrate adequate marrow hemopoietic function as defined below:WBC>3.0×109/L,ANC>1.5×109/L,HGB>90g/L,PLT>80×109/L
  * Demonstrate adequate organ function as defined below: cardiac function grade 0-2（NYHA）；SpO2>88%( natural state)；ALT<3UNL，TBil<2ULN; SCr>60ml/min/m2
  * Having at least one measurable lesions
  * Sign the Informed consent

Exclusion Criteria:

* • The pathological diagnosis was T-cell lymphoma.

  * systemic lymphoma involved CNS
  * Pre-existing uncontrolled active infection
  * Acute myocardial infarction or unstable angina within 6 months; Uncontrolled hypertension and arrhythmia
  * Active bleeding
  * Allergic to any component of the investigational product.
  * Subjects who are suspected to be unable to comply with the study protocol
  * Pregnancy or active lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate | The ORR will be evaluated at 82 days from the POR treatment, which means after 4 cycles and each cycle is 21 days
  ORR is defined as the proportion of patients with a best response of CR, CRu or PR

SECONDARY OUTCOMES:
overall response rate | The ORR will be evaluated at 126 days from date of signing the informed consent , which means after 6 cycles and each cycle is 21 days
  ORR is defined as the proportion of patients with a best response of CR, CRu or PR
complete response rate | The ORR will be evaluated at 82 days from the POR treatment, which means after 4 cycles and each cycle is 21 days
  CR is defined as the proportion of patients with a best response of CR or CRu
2 years progression-free survival | From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow-up without relapsing
2 years overall survival | From date of signing the informed consent until the date of death from any cause, whichever came first, assessed up to 2 years
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow-up alive
The occurrence of adverse events and serious adverse events | during follow-up, up to 2 years
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing TianTan Hospital, Beijing, Beijing Municipality
  - Sanbo Brain Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality